CLINICAL TRIAL: NCT05975515
Title: Effect of Soft Tissue Volume on Midfacial Gingival Margin Alterations Following Immediate Implant Placement in the Esthetic Zone: A 1-Year Randomized Clinical and Volumetric Trial
Brief Title: Midfacial Gingival Margin Changes Following Immediate Implants.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Aboulfettouh, Dr. Ahmed Ibrahim AboulFettouh, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PER 2612
Record Dates: First submitted 2023-07-27; First posted 2023-08-04 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Customized Healing Abutment Bone Grafts Connective Tissue Graft Immediate Implant Placement
MeSH Terms: interventions — Bone Transplantation

STUDY DESIGN:
Intervention Model Description: Randomized controlled clinical trial, parallel groups, three-arm, superiority trial with 1:1:1 allocation ratio.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- immediate implant placement with bone grafts till crest (Active Comparator): Group1 (control group): immediate implant placement with bone grafts till crest and customized healing abutment.
  Interventions: Procedure: Connective tissue graft /Bone graft/ Customized HA
- immediate implant placement with customized healing abutment (Experimental): Group 2 (intervention 1 group): Immediate implant placement with CTG and customized healing abutment.
  Interventions: Procedure: Connective tissue graft /Bone graft/ Customized HA
- immediate implant placement with CTG and customized healing abutment. (Experimental): Group 3 (intervention 2 group): immediate implant placement with customized healing abutment
  Interventions: Procedure: Connective tissue graft /Bone graft/ Customized HA

INTERVENTIONS:
Procedure: Connective tissue graft /Bone graft/ Customized HA — Soft tissue management and augmentation
  Other Names: Customized Healing abutment

SUMMARY:
Dimensional changes, including the loss of labial soft tissues and midfacial gingival recession, seem to be inevitable following immediate placement. The clinical relevance of this study is proposing a treatment modality namely customized healing abutment with immediate implant placement that is proposed to minimize and control midfacial gingival recession and support buccal soft tissue contour, and maintain long term stability of these tissue, which might enhance the esthetics

DETAILED DESCRIPTION:
Tooth extraction is followed by ridge alteration and soft tissue collapse and recession. Different strategies were proposed to limit this collapse however, the ability of these techniques to mimic the original soft tissue level and to maintain long term stability is unclear (Slagter et al., 2014). Using customized contoured healing abutments at the time of immediate implant placement is a treatment modality to improve esthetics by maintaining the soft tissue level and contour (Ruales-Carrera et al, 2019, Perez et al, 2020). Using connective tissue grafts has been suggested to enhance and maintain soft tissue stability, however, the effect of the combined procedures for maintenance of the soft tissue morphology compared to customized healing abutments alone remains unclear (Atieh et al, 2019).

ELIGIBILITY:
Inclusion Criteria:

* Patient-related criteria:

  * Adults at or above the age of 18.
  * Non-restorable maxillary anterior or premolar tooth requiring extraction and needed an implant placing therapy.
  * The failing tooth will have adjacent and opposing natural teeth.
  * Sufficient mesial-distal and interocclusal space for placement of the implant and definitive restoration.
  * Able to tolerate surgical periodontal procedures.
  * Good oral hygiene.
  * Compliance with the maintenance program.
  * Provide informed consent.
  * Accepts the one-year follow-up period.

Teeth related criteria:

* Intact thick biotype gingival tissue with at least 2mm band of keratinized tissue.
* Intact socket wall before the extraction, buccal bone thickness ≤1mm assessed by CBCT.
* Sufficient apical bone to place an immediate implant with minimum primary stability of 30Ncm

Exclusion Criteria:

* Patients diagnosed with periodontal diseases.
* Current or previous smokers.
* Pregnant and lactating females.
* Patients with medical conditions that would compromise the surgical procedures; uncontrolled diabetes mellitus, taking IV Bis-phosphonates for treatment of osteoporosis.
* Patients with active infection related at the site of implant/bone graft placement.
* Patients with parafunctional habits

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2022-01-13 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Midfacial Gingival Margin Changes | 12 months
  will be assessed by measuring the distance between level of soft tissues at mid-facial gingival level of the implant site and a reference line, which connected the facial soft tissue level of the adjacent teeth, at baseline, 3, 6 and 12 months of follow up.

SECONDARY OUTCOMES:
Bone labial to the implant | 12 months
  Two CBCT scans will be done, primary (preoperative) scan and secondary (Postoperative) scan 12 months after, using Cranex ® SOREDEX, Finland.
Volumetric analysis of buccal contour&Total Volume | 12 months
  To evaluate tissue volume changes in the buccal soft tissue contour in comparison to the original ones, at 2,4 and 6 mm from the pre-operative gingival margin, at 3, 6 and 12 months and will be compared to the presurgical scanned casts

CONTACTS AND LOCATIONS:
Locations (1):
- IDCE, Cairo, Egypt

REFERENCES:
- [Derived] Fettouh AIA, Ghallab NA, Ghaffar KA, Elarab AE, Abdel-Aziz NG, Mina NA, Shemais NM, Dahab OA. Effect of soft tissue volume on midfacial gingival margin alterations following immediate implant placement in the esthetic zone: a 1-year randomized clinical and volumetric trial. BMC Oral Health. 2024 Oct 19;24(1):1256. doi: 10.1186/s12903-024-04845-y. PMID 39427143